CLINICAL TRIAL: NCT04856033
Title: A Phase 3 Clinical Trial on Transcendental Meditation and Posttraumatic Stress Disorder, Suicide, and Substance Use in Veterans
Brief Title: Transcendental Meditation and PTSD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: David Lynch Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DLF2021
Record Dates: First submitted 2021-04-16; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Ptsd; Depressive Symptoms; Suicidal Ideation; Alcohol Use, Unspecified
Keywords: Ptsd; Veterans; Meditation; Suicidal ideation; Randomized Controlled Trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Suicidal Ideation; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: 2 group RCT
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TM (Experimental): Transcendental Mediation
  Interventions: Behavioral: TM
- PCT (Active Comparator): Present Centered Therapy
  Interventions: Behavioral: PCT

INTERVENTIONS:
Behavioral: TM — Transcendental Meditation instruction, 12-sessions over 3-4 months with monthly follow-up
  Arms: TM
Behavioral: PCT — Present Centered Therapy, 12-sessions over 3-4 months with monthly follow-up
  Arms: PCT

SUMMARY:
This paper describes the rationale and design of a Phase 3 RCT comparing Transcendental Meditation to Present Centered Therapy for posttraumatic stress disorder (PTSD), suicidal ideation, alcohol use, and depressive symptoms in Veterans. In this multisite trial, 450 Veterans meeting Diagnostic and Statistical Manual-5 (DSM-5) criteria for PTSD will be recruited from nine VA and academic medical center sites across the U.S. Study outcomes include changes in PTSD diagnosis and symptom severity (primary), suicidal ideation, alcohol use, and depressive symptoms. Participation includes baseline testing and post-treatment assessments at 12, 24, and 36-weeks. During each assessment visit, Veterans will complete diagnostic interviews, including the Clinician-Administered PTSD Scale for DSM-5 and the Alcohol Timeline Followback, as well as validated self-report measures. Cost-effectiveness of the treatments will be measured using intervention and healthcare costs, the proportion with PTSD diagnosis removed, and Quality-Adjusted Life Years. Finally, single-site substudies will examine pre-to-post-treatment changes in PTSD biomarkers and on magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Background: The evidence supporting the Transcendental Meditation (TM) technique as a treatment for posttraumatic stress disorder (PTSD) has advanced considerably in the past decade. With a recent randomized controlled trial (RCT) suggesting statistical superiority to active control treatments for PTSD (e.g., Present Centered Therapy [PCT]) and noninferiority to first-line PTSD psychotherapies, additional research evaluating the benefits and cost-effectiveness of TM for PTSD among Veterans is needed.

Methods and design: This paper describes the rationale and design of a Phase 3 RCT comparing TM to PCT for PTSD in Veterans. In this multisite trial, 450 Veterans meeting DSM-5 criteria for PTSD will be recruited from nine VA and academic medical center sites across the U.S. Study outcomes include changes in PTSD diagnosis and symptom severity (primary), suicidal ideation, alcohol use, and depressive symptoms. Participation includes baseline testing and post-treatment assessments at 12, 24, and 36-weeks. During each assessment visit, Veterans will complete diagnostic interviews, including the Clinician-Administered PTSD Scale for DSM-5 and the Alcohol Timeline Followback, as well as validated self-report measures. Cost-effectiveness of the treatments will be measured using intervention and healthcare costs, the proportion with PTSD diagnosis removed, and Quality-Adjusted Life Years. Finally, single-site substudies will examine pre-to-post-treatment changes in PTSD biomarkers and on magnetic resonance imaging (MRI).

Discussion: Despite progress in PTSD treatments, new evidence-based treatments are still needed for Veterans who drop-out of or respond poorly to existing trauma-focused psychotherapies and that may assist Veterans with common PTSD-comorbidities such as depression, suicidal ideation, and substance use. This multisite trial seeks to advance the science and potential application of TM as a treatment for PTSD in Veterans.

ELIGIBILITY:
Inclusion Criteria:

1. Current diagnosis of PTSD from medical record or CAPS-5 interview
2. A symptom severity score≥33 on the CAPS-5 indicating clinically significant PTSD symptoms
3. Three or more months since trauma
4. Agreement to not receive other psychotherapy or meditation for PTSD during the active treatment or follow-up period. Psychotherapy for other problems will be allowed.
5. If being treated with psychoactive medications, a stable regimen (no change in drugs or dose) for at least 2 months before enrollment
6. Age: 18 years or older
7. Language: English literate

Exclusion Criteria:

1. Prior training with TM or treatment with PCT in the past year
2. Currently untreated psychotic symptoms or mania symptoms from chart review or self-report
3. Moderate or greater cognitive impairment indicated by chart diagnosis or observable cognitive difficulties
4. Acute severe symptoms (such as imminent suicidal risk) that will likely require active treatment intervention (such as medication changes) within the course of the study
5. Psychiatric hospitalization in the previous six months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
PTSD diagnosis and symptoms | Baseline, immediately after the intervention, 12-weeks after the intervention, 24-weeks after the intervention
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) changes in PTSD diagnosis and symptom severity. Scores range from 0-80 with higher scores=higher PTSD symptoms

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, immediately after the intervention, 12-weeks after the intervention, 24-weeks after the intervention
  Patient Health Questionnaire-9 (PHQ-9) changes, range=0-27, higher scores=higher depressive symptoms
Alcohol use | Baseline, immediately after the intervention, 12-weeks after the intervention, 24-weeks after the intervention
  Timeline Followback changes
Suicidal ideation | Baseline, immediately after the intervention, 12-weeks after the intervention, 24-weeks after the intervention
  Columbia-Suicide Severity Rating Scale (C-SSRS), range 0-25 with higher scores=greater suicidal ideation intensity

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rutledge, PhD, Principal Investigator — VA San Diego

IPD SHARING:
Plan to Share IPD: No